CLINICAL TRIAL: NCT02579356
Title: A Randomized, Open-label, Multiple-dose, Crossover Study to Evaluate the Drug-drug Interaction Between Telmisartan and Atorvastatin in Healthy Male Volunteers
Brief Title: To Evaluate the Drug-drug Interaction Between Telmisartan and Atorvastatin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SI-1307
Record Dates: First submitted 2015-10-13; First posted 2015-10-19 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Diseases of the Circulatory System; Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Telmisartan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part1-A (Experimental): The Part1-A of groups take Telmisartan once a day for 6 days in period 1. After wash-out period, they take Telmisartan and Atorvastatin once a day for 6 days in period 2.
  Interventions: Drug: Telmisartan; Drug: Atorvastatin
- Part1-B (Experimental): The Part1-B of groups take Telmisartan and Atorvastatin once a day for 6 days in period 1. After wash-out period, they take Telmisartan once a day for 6 days in period 2.
  Interventions: Drug: Telmisartan; Drug: Atorvastatin
- Part2-A (Experimental): The Part2-A of groups take Atorvastatin once a day for 6 days in period 1. After wash-out period, they take Telmisartan and Atorvastatin once a day for 6 days in period 2.
  Interventions: Drug: Telmisartan; Drug: Atorvastatin
- Part2-B (Experimental): The Part2-B of groups take Telmisartan and Atorvastatin once a day for 6 days in period 1. After wash-out period, they take Atorvastatin once a day for 6 days in period 2.
  Interventions: Drug: Telmisartan; Drug: Atorvastatin

INTERVENTIONS:
Drug: Telmisartan
Drug: Atorvastatin

SUMMARY:
The study design was composed of 2 parts, 2-way crossover and multiple-dose. There are having 2 groups in each part that have divided period 1 and period 2, and wash-out period is 16 days between periods. Each group is taking Telmisartan (80mg) and/or Atorvastatin (80mg) once a day for 6 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 19 and 55 years
* Subjects who don't have congenital or chronic diseases and have no abnormal medical examination results within 3 years
* Healthy Subjects (no clinically relevant findings in any of the investigations of the pre-examination) as judged by the investigator
* Subjects who signed and dated in informed consent form indicating that the subject has decided to participate in the study after being informed of all pertinent aspects of the study
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Any condition possibly affecting drug absorption, distribution, metabolism, and excretion (e.g. gastrectomy)
* Twofold or more than upper limit of normal range in laboratory test for ALT or AST
* Participating in other clinical trial study within 2 month preceding the first dose of investigational product
* History of significant alcohol abuse or drug abuse within one year prior to the screening
* Whole blood donation within 2 months prior to dosing, or apheresis donation within 1 month prior to dosing
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study
* Unwilling or unable to comply with the lifestyle guidelines described in this protocol
* Subjects who are inadequate for this study to participate judged by investigator

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
AUCt(0-24) | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)
Css,max | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)

SECONDARY OUTCOMES:
Css,min | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)
Css,av | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)
Tss,max | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)
t1/2 | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)
CL/F | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)
Vd/F | First, fourth, fifth, and sixth day. At 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose in sixth day. (15 times)

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk National University Hospital, Seoul, South Korea